CLINICAL TRIAL: NCT06264557
Title: A Multicenter, Prospective, Comparative, Randomized, Independent Rater-blind, Superiority Clinical Trial to Compare the Safety and Efficacy of the Cognitive Therapy Software 'SUPERBRAIN DEX' With a Control Group for Patients With MCI
Brief Title: Cognitive Therapy Software for Improving Cognitive Function for Patients With Mild Cognitive Impairment
Acronym: SB-DEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rowan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RW-MCI-01; ROWAN (Other: ROWAN)
Record Dates: First submitted 2024-02-08; First posted 2024-02-20 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Mild Cognitive Impairment; MCI
Keywords: SUPERBRAIN; SUPERBRAIN DEX; DEX; MCI; Digital Therapeutics
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): Device : SB-100
  Cognitive training will be conducted once a day, and it will take 15 to 30 minutes.
  It consists of cognitive training and educational videos.
  Interventions: Device: SB-100
- Contol group (Other): Educational book : book of education on daily rules for preventing dementia
  Interventions: Other: Educational book

INTERVENTIONS:
Device: SB-100 — Cognitive training will be conducted once a day, and it will take 15 to 30 minutes.
  It consists of cognitive training and educational videos.
  Arms: Treatment group
Other: Educational book — Book of education on daily rules for preventing dementia
  Arms: Contol group

SUMMARY:
Cognitive therapy software for improving cognitive function for patients with mild cognitive impairment

DETAILED DESCRIPTION:
A multicenter, prospective, comparative, randomized, independent rater-blind, superiority, pivotal clinical trial to compare the safety and efficacy of the Cognitive therapy software 'SUPERBRAIN DEX' for improving cognitive function with a control group for patients with mild cognitive impairment

ELIGIBILITY:
Inclusion Criteria:

1. 50 - 85years old
2. Those who meet all of the National Institute on Aging-Alzheimer's Association (NIA-AA) key clinical criteria below that may suspect mild cognitive impairment caused by Alzheimer's disease as of the screening date

   * Concern of the subject or guardian about the deterioration of cognitive function compared to before
   * More than one cognitive impairment
   * Maintaining the independence of overall daily life functions
   * It's not dementia
3. In at least one of the following neuropsychological tests conducted within one year of the screening date, the delayed recall score in the memory area was 'average -1' according to the standard score table corrected for education level and age.

   * Seoul Neuropsychological Screening Battery 2nd edition (SNSB-II)
   * Korean version of Consortium to Establish a Registry for Alzheimer's Disease (CERAD-K)
   * Literacy Independent Cognitive Assessment (LICA)
4. A person whose Korea-Mini Mental State Examination-2 (K-MMSE-2) score corresponds to "Average-1.5 standard deviation or higher" according to the standard score table corrected for education level and age as of the screening date
5. Those with a Global Clinical Dementia Rating (CDR) score of 0.5 and a memory item score of 0.5 or 1 as of the screening date
6. A person who has a guardian in regular contact with the subject

   * Defined to be able to support subjects during the clinical trial (compliance supervision and subject status reporting) and spend at least 8 hours per week with subjects
7. A person who is taking drugs (donepezil, galantamine, ribastigmine, memantine) for the purpose of improving cognitive function is taking drugs stably for at least 12 weeks as of the screening date
8. Those who have no difficulty using tablet PCs
9. A person who voluntarily decides to participate in this clinical trial and agrees to the subject's explanation and consent in writing
10. Those who are willing to comply with the clinical trial plan

Exclusion Criteria:

1. Those diagnosed with dementia (including Alzheimer's disease, vascular dementia, infections of the central nervous system (e.g., Human Immunodeficiency Virus (HIV), syphilis, etc.), Creutzfeld-Jacob disease (Creutzfeld-Jacob disease), Pick disease, Huntington's disease, Parkinson's disease, etc.) as of the screening date
2. Those who have a history of diagnosing significant neurological diseases affecting cognitive function within one year of the screening date (e.g., stroke, multiple sclerosis, severe head trauma with loss of consciousness, normal cerebral hydrocephalus, epilepsy, brain tumors, cerebral infarction, spinal cord infarction or central nervous system infection)
3. Based on the screening date, major depressive disorder, bipolar disorder, schizophrenia, A person diagnosed with a serious mental illness such as drug addiction and alcoholism
4. Laboratory and/or vital signs tests as of the date of screening, any of the following

   * Those diagnosed with infectious or metabolic diseases that may cause cognitive decline in the subject (e.g., hypothyroidism, vitamin B12 deficiency, folate deficiency, neurotoxin, HIV)
   * Those with liver dysfunction (AST, ALT ≥ 3x upper limit of normal range) and/or renal dysfunction (serum creatinine ≥ 2x upper limit of normal range)
   * Those with uncontrolled hypertension (SBP > 180 mmHg) and/or diabetes (HbA1c > 11%)
5. Those who have severe or unstable cardiovascular disease (e.g., myocardial infarction, unstable angina, class III or IV heart failure by classification of the New York Heart Association (NYHA) within 24 weeks of the screening date)
6. Where the tester determines that he/she has a medical condition that may interfere with the completion of the clinical trial due to a serious or unstable physical condition (e.g., a history of malignant tumors within five years of the screening date (e.g., basal cell cancer and squamous cell carcinoma of the skin considered to have been completely resected and cured, cervical intraepithelial carcinoma, non-transparent prostate cancer, acute and severe asthma, active peptic ulcers, etc.)
7. If you can't walk, A person who can move using walking aids (e.g. walkers, canes, wheelchairs, etc.)
8. an illiterate patient who is unschooled (defined as unadmitted to a regular school)
9. Where the tester determines that a person does not have sufficient vision, hearing, language skills, motor skills, and comprehension to follow the examination procedures related to clinical trials
10. a person who is pregnant or nursing
11. For women of childbearing age, who do not agree with the medically permitted contraceptive method during the clinical trial

    * Hormonal contraception, intrauterine device (IUD) or intrauterine system (IUS), oviduct ligation, double blocking (male condom, female condom, cervical cap, a combination of contraceptive septum, contraceptive sponge-like blocking methods), a single blocking method with a combination of an alveolar agent
12. Those who are currently participating in other clinical trials or who have participated in other clinical trials within 90 days of screening
13. Other, ethical or clinical trial outcomes may be impacted and deemed inappropriate by the tester

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-03-13 (Actual); Study Completion 2025-06-02 (Actual)

PRIMARY OUTCOMES:
K-RBANS | Baseline, 16 weeks after treatment
  The closer the total score of 160 points, the worse the cognitive state is, and the closer it is to 40, the worse the cognitive state is

SECONDARY OUTCOMES:
K-RBANS | Baseline, 8 weeks after treatment
  The closer the total score of 160 points, the worse the cognitive state is, and the closer it is to 40, the worse the cognitive state is
K-MMSE-2 | Baseline, 8 weeks after treatment, and 16 weeks after treatment
  Total scores range from 0 to 30, with lower scores indicating more worsening.
CDR-SB | Baseline, 8 weeks after treatment, and 16 weeks after treatment
  The closer to CDR 0 grade, the more normal the cognitive state, and the closer to CDR 3 grade, the worse the cognitive state.
K-IADL | Baseline, 8 weeks after treatment, and 16 weeks after treatment
  It consists of a total of 11 items (0-3 points), and the score is calculated by dividing the total score by the number of corresponding items, and the closer it is to 3, the worse the cognitive state is.
PRMQ | Baseline, 8 weeks after treatment, and 16 weeks after treatment
  The closer to the lowest 16 points, the normal memory ability, and the closer to the total score of 80 points, the worse the memory ability.
GDS-15 | Baseline, 8 weeks after treatment, and 16 weeks after treatment
  The closer it is to 0, the less depressed it is, and the closer it is to the total score of 15, the more depressed it is.
QOL-AD | Baseline, 8 weeks after treatment, and 16 weeks after treatment
  The closer the total score of 52 points, the higher the quality of life, and the closer the minimum score of 13 points, the lower the quality of life.
ADAS-Cog14 | Baseline, 16 weeks after treatment
  Total scores range from 0 to 90, with higher scores indicating more worsening.

CONTACTS AND LOCATIONS:
Locations (12):
- South Korea (12):
  - Hanyang University Guri Hospital, Guri-si, Gyeonggi-do
  - Inje University Haeundae Paik Hospital, Busan
  - Inha University Hospital, Incheon
  - Gachon University Gil Medical Center, Incheon
  - Chonnam National University Hospital, Kwangju
  - Ewha Womans University Seoul Hospital, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Koera University Guro Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Ajou University Hospital, Suwon
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon

IPD SHARING:
Plan to Share IPD: No